CLINICAL TRIAL: NCT04293952
Title: Comparison of BRACE(Balance, Resistance, Aerobic, and Cognitive Exercises) and BRE (Balance Resistance Exercises) on Fall Risk Reduction in Elderly
Brief Title: Comparison of (Balance, Resistance, Aerobic and Cognitive Exercises) & (Balance Resistance Exercise)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/20/2010 Ayesha Batool
Record Dates: First submitted 2020-03-01; First posted 2020-03-03 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Elderly Population

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRACE group (Experimental): BRACE include combination of exercises including, Balance, Resistance, Aerobic, Cognition Exercises.
  Interventions: Other: Balance, Resistance, Aerobic, Cognition Exercises (BRACE)
- BRE group (Active Comparator): this group include Balance Resistance Exercises Stretching Range Of Motion exercises Ankle flexion Ankle extension Knee flexion Knee extension Hip flexion Hip extension Hip adduction Hip abduction
  Interventions: Other: Balance Resistance Exercise (BRE)

INTERVENTIONS:
Other: Balance, Resistance, Aerobic, Cognition Exercises (BRACE) — BRACE is a combination of different exercises including Balance, Resistance, Aerobic, Cognition for fall risk reduction and to mobility in the elderly.
  Arms: BRACE group
Other: Balance Resistance Exercise (BRE) — this is the simple conventional treatment for the elderly in balance problems including warm-up, resistance exercises and cool-down exercises.
  Arms: BRE group

SUMMARY:
In the elderly risk of fall increased due to impaired balance and gait, cognitive impairment, sensory defects and reduced muscle strength. In this research, the aim of the study is to compare the effect of BRACE (balance, resistance, aerobic exercises and cognitive exercises) and BRE (balance resistance Exercises) on fall risk and mobility level in the elderly population. Randomized control trial study of 6 weeks follows up. The sample size is 40. The patients will be randomly divided into two groups: BRACE and BRE. The patients will get a supervised protocol for 3 days per week for 3 to 9 week. The measurement will be taken at baseline, after 3, 6 and 9 weeks. The study duration is of 8 months. Sampling technique will be purposive sampling and random assignment through the sealed envelope method. Individuals of age above 60 years, either gender with Berg balance score 20-40, MMSE will be included. Individuals with Musculoskeletal conditions (fractures, severe arthritis grade iii and i), Neurological conditions like Epilepsy, Parkinson and Other systemic diseases or co-morbidities will be excluded. Assessment tools will be MMSE, Berg balance scale, TUG, 6 minutes walk test. Data will be analyzed through the Statistical Package for Social Sciences (SPSS) 20.

DETAILED DESCRIPTION:
In terms of morbidity and mortality fall is a major concern in older adults. Fall is defined as unintentional contact with the ground. In 1988 defined fall as "an event in which a person rest unintentionally on the ground or lower surface". There are many reasons for fall which can be intrinsic or extrinsic. The risk factors of fall can be ageing (e.g. cognitive impairment, poor balance or low vision), nutritional (vitamin D and calcium deficiency), medication (sedatives, antidepressants etc), environmental factors (improper shoes, poor lightning and unsafe stairs) and lack of exercise.

The most common mechanism of injury in the elderly population is falling about 30%-50% of falls in the elderly result in minor injuries, including bruises, abrasions, and lacerations, but an estimated 10% of all falls in seniors cause major injuries, including intracranial injuries and fractures. One per cent of all falls in this population result in hip fractures, which pose a significant risk for post-fall morbidity and mortality.

A case series was conducted at Shifa Tamer-e-Millat University Islamabad from January-July 2016. Sixteen adults more than 60 years age (07 males and 09 females) were recruited through convenient sampling. The specified Wii fit plus training was provided to all patients and the games included the Soccer heading, Ski slalom, table tilt and yoga. The Wii fit training improves the balance and reduces the fall risk in the older population.

A study was conducted to evaluate the effects of virtual reality and strength training on the balance, fear of falling and handgrip strength of older women with a history of falls. Balance training consisting of virtual reality and strengthening exercises proved to be an effective tool to reduce the fear of falling and to improve the mobility of elderly female fallers and may be an acceptable treatment for the prevention of falls and balance recovery.

Older adults are prone to fall due to ageing. Mostly older adults aged 60 and above fall due to cognitive impairment, balance problems and physiological functioning. Many studies reported that prevention of fall is possible by adopting a healthy lifestyle, environmental modification, exercise and education. Exercise plays a very important role in fall prevention e.g exercise and tai chi training target balance, flexibility and strength can reduce fall and harm related to fall. Although it does not show a marked difference enjoyable exercise program training is beneficial to achieve healthy outcomes.

In the last few years, several journals had been published specifically on balance training exercises, resistance exercises and aerobic exercises separately. A new tool has been designed for fall risk reduction and to mobility in elderly is BRACE (Balance, Resistance, Aerobic, Cognition Exercises).

A randomized control trial was conducted to compare the effects of S-BRACE (Balance, Resistance, Aerobic, Cognition Exercises) versus conventional therapy on functional balance, mobility and fall risk reduction in elderly with moderate fall risk. It is concluded supervised BRACE training has a better outcome in improving dynamic balance, mobility and risk of fall reduction. Cognitive improvement was observed in both groups.

However, investigation on BRACE protocol is rare in literature. My aim is to compare the effect of BRACE protocol with BRE protocol on mobility and fall risk reduction in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Berg balance score 20-40
* Mini-mental state examination not less than 23

Exclusion Criteria:

* Musculoskeletal conditions (fractures, severe arthritis grade iii and iv)
* Neurological conditions like Epilepsy, Parkinson,
* Alzheimer's, Impaired cognition
* Other systemic diseases or co-morbidities

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | week 9
  changes from the baseline, Berg balance scale (BBS) is used for assessment of balance and fall risk, Higher scores on the BBS indicate greater independence and better ability to balance. In contrast, lower scores indicate a greater fall risk Items DESCRIPTION SCORE (0-4) Sitting to standing, Standing unsupported, Sitting unsupported, Standing to sitting, Transfers , Standing with eyes closed , Standing with feet together, Reaching forward with outstretched arm, Retrieving object from floor, Turning to look behind, Turning 360 degrees, Placing alternate foot on stool, Standing with one foot in front, Standing on one foot, TOTAL __/56
timed up and go test (TUG) | week 9
  changes from the baseline, Timed up and go test is used for the assessment of falls risk among the elderly population. The Timed "Up and Go" (TUG) Test measures, in seconds, the time is taken by an individual to stand up from a standard armchair (approximate seat height of 46 cm, arm height 65 cm), walk a distance of 3 meters (approximately 10 feet), turn, walk back to the chair, and sit down. Normal healthy elderly usually complete the task in 10 seconds or less. Very frail or weak elderly with poor mobility may take 2 minutes or more. Clinical guide: <10 seconds = normal <20 seconds = good mobility, can go out alone, mobile without a gait aid <30 seconds = problems, cannot go outside alone, requires a gait aid A score of more than or equal to 14 seconds has been shown to indicate a high risk of falls.
6 minute walk test | week 9
  The object of this test is to walk as far as possible for 6 minutes. the patient will walk back and forth in this hallway. Six minutes is a long time to walk, so the patient will be exerting. he will probably get out of breath or become exhausted. patients are permitted to slow down, to stop, and to rest as necessary. he may lean against the wall while resting, but resume walking as soon as patients are able. the patient will be walking back and forth around the cones. the patient should pivot briskly around the cones and continue back the other way without hesitation Predictive equation for males: 6 Minute Walk Distance (m) = 867 - (5.71 age, yrs) + (1.03 height, cm) Predictive equation for females: 6 Minute Walk Distance(m) = 525 - (2.86 age, yrs) + (2.71 height, cm) - (6.22 BMI).

SECONDARY OUTCOMES:
Mini mental state examination | day 1
  The Mini-Mental State Exam (MMSE) is a widely used test of cognitive function among the elderly; it includes tests of orientation, attention, memory, language and visual-spatial skills. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Nawaz Malik, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halvarsson A, Franzen E, Stahle A. Balance training with multi-task exercises improves fall-related self-efficacy, gait, balance performance and physical function in older adults with osteoporosis: a randomized controlled trial. Clin Rehabil. 2015 Apr;29(4):365-75. doi: 10.1177/0269215514544983. Epub 2014 Aug 20. PMID 25142277
- [Background] Afridi A, Malik AN, Ali S, Amjad I. Effect of balance training in older adults using Wii fit plus. J Pak Med Assoc. 2018 Mar;68(3):480-483. PMID 29540893
- [Background] Prata MG, Scheicher ME. Effects of strength and balance training on the mobility, fear of falling and grip strength of elderly female fallers. J Bodyw Mov Ther. 2015 Oct;19(4):646-50. doi: 10.1016/j.jbmt.2014.11.013. Epub 2014 Dec 5. PMID 26592222
- [Background] Zhuang J, Huang L, Wu Y, Zhang Y. The effectiveness of a combined exercise intervention on physical fitness factors related to falls in community-dwelling older adults. Clin Interv Aging. 2014;9:131-40. doi: 10.2147/CIA.S56682. Epub 2014 Jan 10. PMID 24453483